CLINICAL TRIAL: NCT04353219
Title: The Effect of Compression Stockings During Training on Running Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 995
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-04

CONDITIONS: Healthy Runners. Compression Stocking and Performance
Keywords: running; performance; compression
MeSH Terms: interventions — Stockings, Compression

STUDY DESIGN:
Intervention Model Description: research group and control group
Who Masked: Participant, Investigator
Masking Description: participant and investigators are not blinded for research groups participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- research group (Experimental): training program with compression stocking
  Interventions: Device: compression stocking
- control group (Active Comparator): training program without compression stocking
  Interventions: Other: control

INTERVENTIONS:
Device: compression stocking — participants will continue their training program as prepared by their coach with compression stocking
  Other Names: compression garments
  Arms: research group
Other: control — participants will continue their training program as prepared by their coach without compression stocking
  Arms: control group

SUMMARY:
Studies that have examined the effects of compression stocking on athlete's performance have been carried out in a single test, i.e., the athlete's was examined during running/riding/jumping with and without the compression stocking.

Yet, using the stocking during all training session and for longer period of time might further enhance the performance. Compression stocking were found to have a positive effect on the athlete' recovery. We hypotheses that if the athlete will train with the stocking on a regular basis and his/her recovery will improve, it will also improve the performance. In addition, the athlete's body may need an adjustment period to use the compression stocking. As such, the advantages of using compression stocking might only be revealed after training with the socks during a period of time and not just performing the tests/competitions with it.

DETAILED DESCRIPTION:
All runners will be examined for: demographical parameters, time of 5 Km run, distance of forward jumping with two leg.

The sample will be divided into 2 research group: research group - all training with compression stocking and control group -training without compression stocking. Both groups will continue their training program for 8 weeks according to their coach. A second examination for the same tests at the end of the 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Runners with at least 3 years of experience and background in competitions (participated in at least 5 competitions participated).
* Train between 4-5 time per week, for minimum of 40 minutes and a minimum of 8 km per training.
* Running minimum 35 km per week.

Exclusion Criteria:

* Runners who practiced in the past with compression stocking.
* Complains of lower limb pains
* Medical history of lower limb or back surgery.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2020-11-27 (Actual)

PRIMARY OUTCOMES:
change from baseline of time running 5 Km | 8 weeks
  time in minutes of running 5 Km
change from baseline of forward two legs jump distance | 8 weeks
  distance of forward jumping in centimeters

SECONDARY OUTCOMES:
change from baseline of average pulse during running | 8 weeks
  heart pulse along the running
change from baseline of maximum pulse during running | 8 weeks
  maximal heart pulse along the running

CONTACTS AND LOCATIONS:
Overall Officials: Gali Dar, PhD, Principal Investigator — Gali Dar, Department of Physical Therapy, University of Haifa
Locations (1):
- Haifa University, Department of PHysical Therapy, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 3 months following study completion

REFERENCES:
- [Background] Ali A, Creasy RH, Edge JA. The effect of graduated compression stockings on running performance. J Strength Cond Res. 2011 May;25(5):1385-92. doi: 10.1519/JSC.0b013e3181d6848e. PMID 21293307